CLINICAL TRIAL: NCT05685992
Title: The Effects and Underlying Mechanisms of Novel Coronavirus Infection on Reproductive Function and Assisted Pregnancy Outcome
Brief Title: Novel Coronavirus Infection and Reproductive Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Bing Yao, Professor, Jinling Hospital, China
Other Study IDs: COVID-19 and reproduction
Record Dates: First submitted 2023-01-12; First posted 2023-01-17 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; Reproductive function; Sustained pregnancy rate
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — serum, seminal plasma, sperm, follicular Fluid, granule cells, embryo culture medium, endometrial tissue, villi and decidual tissue if abortion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infertile couples infected or not infected with COVID-19: Infertile couples infected or not infected with COVID-19 were included.This is an observational study with no interventions.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This study aims to observe the impact of COVID-19 infection on the reproductive function and assisted pregnancy outcome of infertile couples undergoing assisted reproductive technology and to determine which factors are related to the clinical pregnancy rate. A multicenter, prospective, observational cohort study was adopted. Infertile couples who met the selection criteria were included in this study, the SAS anxiety self-rating scale was filled out, the basic situation was observed, and blood samples and related tissues were collected for testing. Relevant reproductive function, laboratory, clinical, and psychological indicators were collected, and the correlation between the above indicators and the outcome of the ART-related pregnancy were analyzed.

DETAILED DESCRIPTION:
In this multicenter, prospective, observational cohort study, we included infertile couples based on inclusion criteria. The couples were asked to fill in the SAS anxiety self-rating scale. Basic information about patients' vaccination status, symptoms related to viral infection, menstruation, sexual desire, and sexual function were obtained. Blood samples of couples were collected on the date of diagnosis, the start date of the fresh cycle during assisted reproductive technology treatment, the day of oocyte retrieval, the day of embryo transfer, the day of 14 days, 35 days after embryo transfer, and the day of 70 days of gestation. Follicular fluid, granulosa cells on the day of oocyte retrieval, and embryo culture fluid on the day of embryo transfer were collected. Blood samples and endometrial tissues were collected five days after oocyte retrieval. Blood samples from the menstrual period, endometrial transformation day, and embryo transfer day of the frozen embryo transfer cycle were also collected. Then C-reactive protein, erythrocyte sedimentation rate, procalcitonin and IL-6, granulocyte-macrophage colony-stimulating factor (GM-CSF), TNF-α, VEGF, and other cytokines and chemokines were determined. In addition, fasting blood glucose, insulin, blood lipids, alpha-function, renin-angiotensinase, I-aldosterone, and other susceptibility indicators to COVID-19 infection were tested. Oxygen saturation, malondialdehyde (MDA), HO-1, and SOD oxidative stress indices of the fingertip pulse were determined. An endometrial receptivity gene chip and proteomics detected endometrial tissue. A panel kit for blood vessel and inflammation indicators detected the abortion decidua tissue. Reproductive function indices AMH, INHB, sex hormones, follicle retrieval rate, Gn days, total Gn, endometrial thickness, the incidence of OHSS, semen quality, oocyte maturation rate, fertilization rate, qualified embryo rate, blastocyst formation rate, and other laboratory indices of both men and women were collected. Assisted pregnancy outcome: clinical pregnancy rate, embryo implantation rate, early abortion rate, ongoing pregnancy rate, and other clinical indicators, as well as psychological indicators such as the SAS anxiety scale, were analyzed to determine the correlation between the above indicators and ART-related pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with infertility

Exclusion Criteria:

* Patients with contraindications to pregnancy or assisted reproductive technology

Ages: 20 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Failure to establish a clinical pregnancy after 12 months of regular unprotected intercourse, or due to impaired fertility of the individual or his or her partner, is termed infertility.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 1 year
  If the fetal sac, fetal bud, and primitive fetal heartbeat are found by vaginal B-ultrasound examination 55-65 days after embryo transfer, the diagnosis of ongoing pregnancy will be made.

SECONDARY OUTCOMES:
Clinical and laboratory indicators related to male and female reproductive function | 1 year
  AMH, INB, sex hormone, follicle output rate, Gn days, total Gn, endometrial thickness on the embryo transfer day, semen quality; Oocyte maturation rate, fertilization rate, high-level embryo rate, blastocyst formation rate
Outcome indicators of assisted pregnancy | 1 year
  Embryo implantation rate, early abortion rate, ongoing pregnancy rate, incidence of OHSS

OTHER OUTCOMES:
Coagulation index | 1 year
  D-dimer
Indicators of susceptibility to COVID-19 infection | 1 year
  blood lipid, blood sugar, insulinand thyroid function
Oxidative stress index | 1 year
  fingertip pulse oxygen saturation
SAS Anxiety Scale | 1 year
  SAS Anxiety Scale

CONTACTS AND LOCATIONS:
Overall Officials: Bing Yao, PHD, Study Chair — Department of Reproductive Medicine, Jinling Hospital; Li Chen, PHD, Study Director — Department of Reproductive Medicine, Jinling Hospital; Xiaojie Huang, PHD, Principal Investigator — Department of Reproductive Medicine, Xuzhou Maternal and Child Health Care Hospital; Jiayi Ding, PHD, Principal Investigator — Department of Reproductive Medicine, Nantong Maternal and Child Health Care Hospital; Qin Sun, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Meiling Li, PHD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Cheng Zhou, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Xi Chen, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Yuming Feng, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Juanjuan Xu, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Haiyan Fu, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Cencen Wang, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Hong Zhang, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Lu Zheng, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Yuxiu Liu, PHD, Principal Investigator — Department of Critical Care Medicine, Jinling Hospital; Xiaofang Tan, MD, Principal Investigator — Department of Reproductive Medicine, Nantong Maternal and Child Health Care Hospital; Yunxia Zhu, MD, Principal Investigator — Department of Reproductive Medicine, Xuzhou Maternal and Child Health Care Hospital; Jueraitetibaike Kadiliya, PHD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital; Zhichan Zou, MD, Principal Investigator — Department of Reproductive Medicine, Jinling Hospital
Locations (3):
- China (3):
  - Department for Reproductive Medicine, Jinling Hospital, Nanjing, Jiangsu
  - Department of Reproductive Medicine, Nantong Maternal and Child Health Care Hospital, Nantong, Jiangsu
  - Department of Reproductive Medicine, Xuzhou Maternal and Child Health Care Hospital, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rodriguez-Morales AJ, Cardona-Ospina JA, Gutierrez-Ocampo E, Villamizar-Pena R, Holguin-Rivera Y, Escalera-Antezana JP, Alvarado-Arnez LE, Bonilla-Aldana DK, Franco-Paredes C, Henao-Martinez AF, Paniz-Mondolfi A, Lagos-Grisales GJ, Ramirez-Vallejo E, Suarez JA, Zambrano LI, Villamil-Gomez WE, Balbin-Ramon GJ, Rabaan AA, Harapan H, Dhama K, Nishiura H, Kataoka H, Ahmad T, Sah R; Latin American Network of Coronavirus Disease 2019-COVID-19 Research (LANCOVID-19). Electronic address: https://www.lancovid.org. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Mar-Apr;34:101623. doi: 10.1016/j.tmaid.2020.101623. Epub 2020 Mar 13. PMID 32179124
- [Background] Chu H, Zhou J, Wong BH, Li C, Chan JF, Cheng ZS, Yang D, Wang D, Lee AC, Li C, Yeung ML, Cai JP, Chan IH, Ho WK, To KK, Zheng BJ, Yao Y, Qin C, Yuen KY. Middle East Respiratory Syndrome Coronavirus Efficiently Infects Human Primary T Lymphocytes and Activates the Extrinsic and Intrinsic Apoptosis Pathways. J Infect Dis. 2016 Mar 15;213(6):904-14. doi: 10.1093/infdis/jiv380. Epub 2015 Jul 22. PMID 26203058
- [Background] Xia W, Shao J, Guo Y, Peng X, Li Z, Hu D. Clinical and CT features in pediatric patients with COVID-19 infection: Different points from adults. Pediatr Pulmonol. 2020 May;55(5):1169-1174. doi: 10.1002/ppul.24718. Epub 2020 Mar 5. PMID 32134205
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Conti P, Ronconi G, Caraffa A, Gallenga CE, Ross R, Frydas I, Kritas SK. Induction of pro-inflammatory cytokines (IL-1 and IL-6) and lung inflammation by Coronavirus-19 (COVI-19 or SARS-CoV-2): anti-inflammatory strategies. J Biol Regul Homeost Agents. 2020 March-April,;34(2):327-331. doi: 10.23812/CONTI-E. PMID 32171193
- [Background] Bobrova L, Kozlovskaya N, Korotchaeva Y, Bobkova I, Kamyshova E, Moiseev S. Microvascular COVID-19 lung vessels obstructive thromboinflammatory syndrome (MicroCLOTS): a new variant of thrombotic microangiopathy? Crit Care Resusc. 2020 Sep;22(3):284. doi: 10.1016/S1441-2772(23)00399-X. No abstract available. PMID 32900338
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Danzi GB, Loffi M, Galeazzi G, Gherbesi E. Acute pulmonary embolism and COVID-19 pneumonia: a random association? Eur Heart J. 2020 May 14;41(19):1858. doi: 10.1093/eurheartj/ehaa254. No abstract available. PMID 32227120
- [Background] Thachil J, Tang N, Gando S, Falanga A, Cattaneo M, Levi M, Clark C, Iba T. ISTH interim guidance on recognition and management of coagulopathy in COVID-19. J Thromb Haemost. 2020 May;18(5):1023-1026. doi: 10.1111/jth.14810. Epub 2020 Apr 27. No abstract available. PMID 32338827
- [Background] Wu M, Ma L, Xue L, Zhu Q, Zhou S, Dai J, Yan W, Zhang J, Wang S. Co-expression of the SARS-CoV-2 entry molecules ACE2 and TMPRSS2 in human ovaries: Identification of cell types and trends with age. Genomics. 2021 Nov;113(6):3449-3460. doi: 10.1016/j.ygeno.2021.08.012. Epub 2021 Aug 18. PMID 34418496
- [Background] Boudry L, Essahib W, Mateizel I, Van de Velde H, De Geyter D, Pierard D, Waelput W, Uvin V, Tournaye H, De Vos M, De Brucker M. Undetectable viral RNA in follicular fluid, cumulus cells, and endometrial tissue samples in SARS-CoV-2-positive women. Fertil Steril. 2022 Apr;117(4):771-780. doi: 10.1016/j.fertnstert.2021.12.032. Epub 2022 Jan 1. PMID 35272846
- [Background] Li K, Chen G, Hou H, Liao Q, Chen J, Bai H, Lee S, Wang C, Li H, Cheng L, Ai J. Analysis of sex hormones and menstruation in COVID-19 women of child-bearing age. Reprod Biomed Online. 2021 Jan;42(1):260-267. doi: 10.1016/j.rbmo.2020.09.020. Epub 2020 Sep 29. PMID 33288478
- [Background] Madendag IC, Madendag Y, Ozdemir AT. COVID-19 disease does not cause ovarian injury in women of reproductive age: an observational before-and-after COVID-19 study. Reprod Biomed Online. 2022 Jul;45(1):153-158. doi: 10.1016/j.rbmo.2022.03.002. Epub 2022 Mar 5. PMID 35523708
- [Background] Henarejos-Castillo I, Sebastian-Leon P, Devesa-Peiro A, Pellicer A, Diaz-Gimeno P. SARS-CoV-2 infection risk assessment in the endometrium: viral infection-related gene expression across the menstrual cycle. Fertil Steril. 2020 Aug;114(2):223-232. doi: 10.1016/j.fertnstert.2020.06.026. Epub 2020 Jun 17. PMID 32641214
- [Background] Youngster M, Avraham S, Yaakov O, Landau Rabbi M, Gat I, Yerushalmi G, Sverdlove R, Baum M, Maman E, Hourvitz A, Kedem A. IVF under COVID-19: treatment outcomes of fresh ART cycles. Hum Reprod. 2022 May 3;37(5):947-953. doi: 10.1093/humrep/deac043. PMID 35212741